CLINICAL TRIAL: NCT03978052
Title: Prevention of Cognitive Decline in ApoE4 Carriers With Subjective Cognitive Decline After EGCG and a Multimodal Intervention
Acronym: (PENSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital del Mar Research Institute (Unknown); Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, Director Neurosciences Research Programme, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IMIM/PENSA
Record Dates: First submitted 2019-05-29; First posted 2019-06-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Cognitive Decline
Keywords: EGCG; Dietary supplement; Personalized medicine; Subjective Cognitive Decline (SCD); Apolipoprotein E4; Lifestyle Risk Reduction; Epigallocatechin gallate; Multimodal lifestyle intervention
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Arm I: EGCG and a multimodal intervention (n=50) Arm II: Placebo EGCG and a multimodal intervention (n=50) Arm III: Healthy lifestyle recommendations (n=50)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind clinical trial (participant, investigator, outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EGCG + multimodal intervention (Experimental): EGCG + multimodal intervention (n=50) EGCG: (Font-UP, Laboratoires Grand Fontaine), a daily dose of 5-6 mg/kg up to 500 mg/day for 12 months
  + multimodal lifestyle personalized intervention
  Interventions: Dietary Supplement: EGCG; Other: Multimodal lifestyle intervention
- Placebo + multimodal intervention (Placebo Comparator): Placebo Font-Up (n=50)
  + multimodal lifestyle personalized intervention
  Interventions: Dietary Supplement: Placebo EGCG; Other: Multimodal lifestyle intervention
- Control (Sham Comparator): Healthy lifestyle recommendations (n=50)
  Interventions: Other: Healthy lifestyle recommendations

INTERVENTIONS:
Dietary Supplement: EGCG — FontUp capsules (100 mg of EGCG each)
  12 months, three to five capsules per day (participant's weight ≤ 50kg: 3 capsules/day; weight >50kg: 5 capsules/day.
  Arms: EGCG + multimodal intervention
Dietary Supplement: Placebo EGCG — Placebo FontUp (same appearance as active).
  12 months, three to five capsules per day (participant's weight ≤ 50kg: 3 capsules/day; weight >50kg: 5 capsules/day.
  Arms: Placebo + multimodal intervention
Other: Healthy lifestyle recommendations — Personalized advice on diet, physical activity, cognitive training, and social stimulation activities.
  Arms: Control
Other: Multimodal lifestyle intervention — * Dietary intervention: personalized dietary recommendations based on MedDiet, 9 individual counseling sessions.
  * Physical activity intervention: Guided gymnasium (aerobic, strength, and balance activities). Minimum one class/week the first 6months, and two classes/week from month 7 to 12). Achieve a physically active lifestyle (10,000 steps/day; individuals living with disability 8,500 steps/day). Achieve moderate physical exercise in older adults (150 to 210 minutes/week or 90 to 150 minutes depending on medical history.
  * Cognitive training: NeuronUP, 3/week, 30 min sessions
  * Psychoeducation: ten 90-minute sessions
  * Social stimulation activities: ten to twelve 90-to-120-minute sessions.
  Arms: EGCG + multimodal intervention; Placebo + multimodal intervention

SUMMARY:
Alzheimer's disease (AD) neuropathology is characterized by deposits of insoluble amyloid β-peptide (Aβ) in extracellular plaques and aggregated tau protein, which is found largely in the intracellular neurofibrillary tangles. Current knowledge, has allowed a shift in the definition of AD from a syndromal to a biological construct, based on biomarkers that are proxies of pathology. However, little is known about mechanisms underlying the disease progression at its early stages. The loss of dendritic spines, the primary locus of excitatory synaptic transmission in the mammalian central nervous may be linked to cognitive and memory impairment in AD: A multimodal lifestyle change intervention (dietary, physical activity and cognition) combined with epigallocatechin gallate (EGCG) will slow down cognitive decline and improve brain connectivity in a population of participants with subjective cognitive decline (SCD). In humans, alterations in functional connectivity (FC) have been observed in early AD stages, subjective cognitive decline (SCD) and mild cognitive impairment (MCI). A hyper-synchronized anterior network and a posterior network characterized by a decrease in FC are the spatial features. These disruptions also seen in AD indicate that FC alterations appear very early in the course of the disease . Experimental research strongly suggests that in order to increase our cerebral reserves, we have to follow a lifestyle that takes into account many factors. Clinical studies provided evidence that individuals with more cerebral reserves are those who have a high level of education, who maintain regular physical activity and who eat in a healthy way. The environmental enrichment (EE) animal models confirmed that the experience plays a key role in increasing brain plasticity phenomena .There is a growing understanding that a valid therapeutic emerging approach in AD is prevention. A large number of modifiable risk factors for AD have been identified in observational studies, many of which do not appear to exert effects through amyloid or tau. This suggests that primary prevention studies focusing on risk reduction and lifestyle modification may offer additional benefits. The therapeutic approach proposed in the present project aims at improving synaptic plasticity and functional connectivity in early stages of AD, and specifically in SCD in the context of a personalized medicine approach that includes a multimodal intervention (nutritional, physical, cognitive and medical) looking at improving person-centered outcomes. In this context the proposed clinical trial design will evaluate the efficacy of EGCG in the context of a personalized medicine approach that includes a multimodal intervention (nutritional, physical, cognitive and medical) looking at improving person-centered outcomes. Early phase I studies in Down syndrome young adults showed that while subjects were under EGCG, improvements in cognition were observed but these vanished when treatment was discontinued. Phase II studies combining EGCG with cognitive training showed improvements in cognitive performance and adaptive functionality but interestingly sustained effects after treatment discontinuation. Observations made in humans are in agreement with preclinical studies showing that EGCG combined with environmental enrichment resulted in an improvement of age-related cognitive decline. These observations are in favor of the option of combining EGCG with a personalized multimodal intervention. The personalized multimodal intervention will take into account medical comorbidities (i.e. metabolic syndrome, T2DM), diet (including nutritional status), physical exercise, and will incorporate cognitive training and a behavioral intervention to aid subject's adherence and empowerment to the intervention proposed. This will be in-line with other clinical studies in AD showing the superiority of multimodal interventions vs. a single life style intervention (i.e. single nutrient, physical activity). Hypothesis: A multimodal lifestyle change intervention (dietary, physical activity and cognition) combined with epigallocatechin gallate (EGCG) will slow down cognitive decline and improve brain connectivity in a population of participants with subjective cognitive decline (SCD).

DETAILED DESCRIPTION:
Study Design: Randomized, double-blind, personalized clinical trial with 150 subjects with subjective cognitive decline (SCD) of both genders, with 3 arms of treatment Duration of the Study: The total duration of the study is expected to be 24 months (subject recruitment, baseline period, treatment period, follow-up, data analysis, and study report).

Primary Objective(s): To evaluate the efficacy of a multimodal intervention (dietary, physical activity, and cognition) combined with epigallocatechin gallate (EGCG) in slowing down cognitive decline.

Secondary Objective(s): 1 To evaluate the safety of the interventions 2 To evaluate several underlying mechanisms that could explain the efficacy of the intervention in preventing the progression of cognitive decline: (i) Changes in brain connectivity, (ii) changes in AD biomarkers, (iii) changes in biomarkers of oxidation/inflammation, (iv) changes in gut microbiota composition and the metabolome derived by the action of microorganisms, v) changes in biological aging predictors.

Target Population: Subjects diagnosed with Subjective Cognitive Decline (SCD) criteria including cognitive performance within normal values (Normal scoring on psychometric evaluation, adjusted for age and education), carriers of the Apolipoprotein E4 allele, recruited either from either the Parc de Salut Mar and its primary care providers, from Barcelona Beta Brain Research Centre or through a web-based system.

Preselection criteria i.Adults aged 60-80 years with a BMI ≥18.5 and <32 kg/m2. ii. Ad-hoc Subjective Cognitive Decline Questionnaire (SCD-Q) item "do you perceive memory or cognitive difficulties?" positive.

iii. Subjects willing to participate and perform all study procedures, including Apolipoprotein E4 genotyping iv. The subject has one informant partner who, in the investigator's judgment has frequent and sufficient contact with the subject to provide accurate information about the subject's cognitive and functional abilities.

Study Arm(s):

1. Arm I: EGCG and multimodal intervention (n=50)
2. Arm II: Placebo EGCG and multimodal intervention (n=50)
3. Arm III: Healthy lifestyle recommendations (n=50) Duration of Patient Participation: The total duration of patient participation is expected to be 17 months. Run-in period (1 month): Basal assessment of cognitive performance (cognitive battery), diet and physical activity, daily living activities (self-reported tests), and mood (self-reported tests at basal assessment and EMA's). Interventions will last 12 months. Follow-up after intervention discontinuation: at least 3 months Treatment: EGCG (Font-UP, laboratories Grand Fontaine), a daily dose of approximately 5-6 mg/kg up to 500 mg/day will be administered to subjects for 12 months or a matched placebo Multimodal intervention (12 months): 1) Social stimulation, ten 90-120 minutes guided group activities; 2) Cognitive training, trice per week, 30-minute sessions; 3) Psychoeducational support groups, 10 sessions, 4) personalized diet 8 sessions, 5) personalized physical activity.

End point: modified Alzheimer Disease Cooperative Study Preclinical Alzheimer Cognitive Composite (ADCS-PACC), including additional tests of executive functions: the PACC-exe.

ELIGIBILITY:
Inclusion Criteria:

i. Meet all selection criteria and no exclusion criteria. ii. Fulfill SCD criteria (Jessen et al. 2014) including cognitive performance within normal values (Normal scoring on psychometric evaluation, adjusted for age and education).

iii. Age between 60 and 80 with a BMI ≥18.5 and <35 kg/m2. iv. Carrying the APOE-ɛ4 allele. v. Participants are willing to participate and perform all study procedures.

Exclusion Criteria:

i. Inability or unwillingness to give written informed consent or communicate with study staff or illiteracy.

ii. Clinically significant unstable psychiatric disorder that may affect cognition (e.g. major depression disorder, schizophrenia, bipolar or psychotic disorder according to DSM-V).

iii. Neurological conditions that may affect cognition or may imply a prodromal stage of neurodegenerative disease other than AD (e.g., cranioencephalic trauma with permanent neurologic effects, epilepsy, multiple sclerosis, previous stroke, extrapyramidal signs at physical exploration, history of brain tumor...).

iv. History or evidence of any medical condition or use of medication that in the opinion of the investigator could affect subjects' safety or interfere with the study assessments (e.g. use of neuroleptic drugs, anticonvulsant medications (except gabapentin and pregabalin for non-seizure indications) corticosteroids or immunosuppressive therapies that may affect inflammatory parameters).

v. Any contraindication to perform brain MRI (e.g. pacemaker, MRI-incompatible aneurysm clips).

vi. Clinically significant abnormalities in laboratory test or MRI scan results at screening unless acceptable by the investigator (e.g. mild/moderate kidney failure, benign tumor that does not require surgical intervention…).

vii. Any medical condition that may affect the study assessments in the opinion of the principal investigators or medical advisors.

viii. Current intake of vitamin supplements, catechins, or products containing EGCG (i.e. TEAVIGO, Mega Green Tea Capsules Life Extension, or Font-UP Grand Fontaine Laboratories) for at least 3 months previous to the screening visit.

ix. History within the last 2 years of treatment for primary or recurrent malignant disease, excluding non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or situ prostate cancer with normal prostate-specific antigen post-treatment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Modified Alzheimer Disease Cooperative Study Preclinical Alzheimer Cognitive Composite (ADCS-PACC) including additional tests of executive functions: the PACC-exe | Screening and 12 months
  Changes in the PACC-exe, that include:
  The Total Recall score from the Free and Cued Selective Reminding Test (FCSRT) (which range from 0-48 words),The Delayed Recall score on the Logical Memory IIa subtest from the Wechsler Memory Scale (which range from 0-25 story units), the Coding Test Total score from the Wechsler Adult Intelligence Scale-Revised (which range from 0-93 symbols), The Montreal Cognitive assessment (MOCA) total score (which range from 0-30 points), and additionally, the Interference score from the Stroop Colour and Word Test (SCWT) and the Five Digit Test. Each of the component change scores is divided by the baseline sample standard deviation of that component, to form standardized z scores. These z scores are summed to form the composite.

SECONDARY OUTCOMES:
Safety outcome of the intervention with EGCG: AEs and SAEs | Baseline, 6 and 12
  evaluated by means of Incidence, nature, severity and causality of adverse events (AEs) and serious adverse events (SAEs)
Safety outcome of the intervention with EGCG: Biomarkers thyroid | Baseline, 6 and 12
  Assessment of thyroid function parameters: both TSH and freeT4 within normal values according to the reference population
Safety outcome of the intervention with EGCG: Biomarkers liver | Baseline, 6 and 12
  Assessment of liver function parameters: ALP and ALT within normal values according to the reference population
Safety outcome of the intervention with EGCG: Biomarkers | Baseline, 6 and 12
  Assessment of renal function parameters: creatinine within normal values according to the reference population
Changes in Functional neuronal connectivity (assessed by a functional magnetic resonance imaging) | Screening and 12 months.
  Changes in Maps of change in connectivity of the Default mode network Changes in Maps of change in connectivity of the Limbic network Changes in Maps of change in connectivity of the Salience network
Changes in structural connectivity networks known to be affected in Alzheimer Disease | Screening and 12 months.
  Changes in Connectivity changes of the parahippocampus/fornix Changes in Connectivity changes of the cingulum/cingulate fiber bundle Changes in connectivity changes of the caudate heads

OTHER OUTCOMES:
Changes in Modified Alzheimer Disease Cooperative Study Preclinical Alzheimer Cognitive Composite (ADCS-PACC) including additional tests of executive functions: the PACC-exe | Screening, 6, 12 and 15 months.
  Changes in the PACC-exe, that include:
  The Total Recall score from the Free and Cued Selective Reminding Test (FCSRT) (which range from 0-48 words),The Delayed Recall score on the Logical Memory IIa subtest from the Wechsler Memory Scale (which range from 0-25 story units), the Coding Test Total score from the Wechsler Adult Intelligence Scale-Revised (which range from 0-93 symbols), The Montreal Cognitive assessment (MOCA) total score (which range from 0-30 points), and additionally, the Interference score from the Stroop Colour and Word Test (SCWT) and the Five Digit Test. Each of the component change scores is divided by the baseline sample standard deviation of that component, to form standardized z scores. These z scores are summed to form the composite.
Changes in the microbiota composition | Baseline, and 12 months.
  For the analysis of microbiota biomarkers our characterization of the microbiome of the samples will include determination of the levels of biodiversity in the samples. Samples will be divided into quartiles in order to label each sample as having low (1st quartile), average (2nd and 3rd quartiles), or high diversity (4th quartile).
Change in the dietary patterns (metabolomics) Plasma samples | Baseline, 6, 12 and 15 months
  Change in the dietary patterns (metabolomics). Plasma, samples will be collected to analyze the corresponding metabolomes (SFCAs, kynurenine pathway...), we will divide samples into quartiles to label each sample as having low (1st quartile), average (2nd and 3rd quartiles), or high diversity (4th quartile)
Change in the dietary patterns (metabolomics) oral fluid | Baseline, 6, 12 and 15 months
  Changes in the dietary patterns (metabolomics) of oral fluid will be collected to analyze the corresponding metabolomes for a better understanding of the complexity of the interrelationship of metabolomics in oral fluid and mental health.
Change in the dietary patterns (metabolomics). urinary samples | Baseline, 6, 12 and 15 months
  Change in the dietary patterns (metabolomics). urinary samples will be collected to analyze the corresponding metabolomes for a better understanding of the complexity of the interrelationship of microbiota, diet, and mental health.
Exploratory | At 6 and 12 months
  Change in metabolomes derived from the treatment compliance after a multimodal lifestyle change intervention. Urinary samples (24h) will be used to identify objective biomarkers of dietary intake and dietary patterns and to assess the degree of adherence to the Mediterranean diet by monitoring the levels of dietary metabolites (i.e. hydroxytyrosol metabolism, biomarkers of alcohol consumption...).
Changes in the semantic verbal fluency | Baseline, 6, 12 and 15 months
  Changes in additional cognitive performance scores of: (i) Semantic verbal fluency, "animals" in one minute. (which range from 0-12 words) higher score is better outcome.
Changes in the Boston Naming Test | Baseline, 6, 12 and 15 months
  Changes in additional cognitive performance scores of: (ii) naming, Boston Naming Test (BNT).: (which range from 0-15 points) higher score is better outcome.
Change in attention and working memory | Baseline, 6, 12 and 15 months
  Changes in additional cognitive performance scores of: (iii) attention and working memory,
Change in the Digit span subtest (WAIS IV) | Baseline, 6, 12 and 15 months
  Changes in additional cognitive performance scores of: (iv) Digit span subtest (WAIS IV) , (which range from 0-16 points)
Changes in the Olfactory function | Baseline, and 12 months
  Changes in the Olfactory function: the University of Pennsylvania Smell Identification Test (UPSIT) is designed to test the function of an individual's olfactory system. It is the gold standard of smell identification tests. Its performance has been related to cognition and it has been widely used as a complementary assessment tool in dementia patients.( which range from 0-40)
Changes in the AD biomarkers | Baseline, and 12 months
  Changes in the AD biomarkers related to neurodegeneration (NfL), neurotoxicity (GFAP),Tau proteins amyloid-β peptides
Changes in biological aging | Baseline and 12 months
  Blood sample will be collected for further analysis on biological age biomarkers assessed by epigenetics (biological ageing). The difference between chronological age and biological age, defined as average age acceleration (Δage), will be used to determine individual aging.
Changes in physical activity/fitness: VREM | Screening, 6, 12 and 15 months
  Changes in physical activity as measured by the Spanish Short Version of the Minnesota Leisure Time Physical Activity Questionnaire (Comellas et al., 2012). It reports energy expenditure during leisure time and allows individuals to be classified into activity categories.
Changes in physical activity/fitness: RAPA | Screening, 6, 12 and 15 months
  Changes in physical activity as measured by the Rapid Assessment of Physical Activity (RAPA). Designed for quickly assessing the level of physical activity of older adults.
Changes in physical activity/fitness: SPPB | Screening, 6, 12 and 15 months
  Changes in physical performance as measured by The Short Physical Performance Battery (SPPB), a validated measure of physical function in older adults. The SPPB represents the sum of results from three component tests of functional relevance: standing balance, 4-meter gait speed (4MGS), and five-repetition sit-to-stand motion (5STS)
Changes in physical activity/fitness: SFT | Screening, 6, 12
  Changes in physical performance as measured by the The Senior Fitness Test battery evaluating balance (flamingo test), lower limb strength (chair stand test), upper limb strength (arm curl test), lower limb flexibility (chair sit-and-reach test), upper limb flexibility (back scratch test), agility (8-foot up-and-go test), speed (brisk walking test) and resistance (6-minute walk test).
Changes in physical activity/fitness: grip strength | Screening, 6, 12 and 15 months
  Changes in physical performance as measured by the grip strength with a dynamometer, which measures the maximum isometric strength of the hand and forearm muscles.
Changes in physical activity/fitness: Fitbit steps | Screening, 6, 12 and 15 months or continuous measures (Fitbit measures and EMAs)
  Changes in physical activity as measured by the number of steps
Changes in physical activity/fitness: Fitbit physical activity | Continuous measure
  Changes in physical activity as measured by the physical activity estimation. Each minute is classified as being sedentary, light, moderate or vigorous activity, based on metabolic equivalent (METs), which are indicators for exercise intensity. After 10 minutes of continuous moderate to intense activity, equivalent for activities at or above 3 METs, such minutes are considered "active minutes".
Changes in physical activity/fitness: Fitbit floors climbed | Continuous measure
  Changes in physical activity as measured by the number of floors climbed
Changes in physical activity/fitness: Fitbit active minutes | Continuous measure
  Changes in physical activity as measured by the number of active minutes
Changes in physical activity/fitness: Fitbit heart rate | Continuous measure
  Changes in physical activity as measured by the heart rate
Changes in quality of sleep: Fitbit sleep | Continuous measure
  Changes in sleep as measured by the sleep duration
Changes in quality of sleep: Pittsburg Sleep Quality Index | Screening, 6, 12 and 15 months
  Changes in sleep measured by the Pittsburg Sleep Quality Index: provides a global index of sleep quality over the previous one-month interval. It is a generic, 19 items self-rated scale designed to measure overall sleep problems
Changes in quality of sleep: Epworth sleepines scale | Screening, 6, 12 and 15 months
  Changes in sleep Epworth sleepiness scale (ESS): The ESS assesses daytime sleepiness. It is a four-grade scale (0, no napping; 3, high likelihood of napping), with eight questions, with a maximum of 24 points; a score >10 is considered to be excessive sleepiness.
Treatment compliance/adherence: EGCG | Screening, 6 and 12 months
  As a biomarker of EGCG ingestion compliance, EGCG will determined in plasma samples by HPLC/MS/MS at 6 and 12 months.
Treatment adherence: Diet | Screening, 6 and 12 months
  Compliance/adherence with diet will be assessed by means of 3-day food diaries
Treatment compliance/adherence: mental health | Screening, 6 and 12 months
  Adherence to mental health interventions will be assessed through means of: (i) monitoring the attendance to the psychoeducational group sessions, (ii) monitoring the attendance to the monthly cognitive stimulation activities, and (iii) monitoring the attendance to the scheduled cognitive training sessions (NeuronUp).
Treatment compliance/adherence: MedDiet-index | Screening, 6 and 12 months
  Compliance/adherence with diet will be assessed by means of the 14-item Mediterranean Diet adherence screener (Martínez-González MA et al. 2012)
Treatment compliance/adherence: Diet MNA | Screening, 6 and 12 months
  Compliance/adherence diet as assessed by the Mini Nutritional Assessment test (MNA), a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. The MNA test is composed of simple measurements and brief questions that can be completed in about 10 min. The sum of the MNA score distinguishes between elderly patients with: 1) adequate nutritional status, MNA > or = 24; 2) protein-calorie malnutrition, MNA < 17; 3) at risk of malnutrition.
Changes in adaptive behaviour: ABAS-2 | Screening, 6, 12 and 15 months
  Changes in adaptive behavior as measured by the Adaptive Behavior Assessment System - Second Edition -ABAS-II- for adults. The ABAS-II tool for adults (ages 16 to 89) includes 5 subscales which assess the individual's competence (in terms of behavior frequency) in 10 different skill areas: communication abilities, community use, functional academics, home living, health and safety, leisure, self-care, self-direction, social interaction and working/labor skills
Changes in Quality of Life: EQ-5D-5L | Screening, 6, 12 and 15 months
  Changes in quality of Life as measured by the EuroQol 5 dimensions 5 levels (EQ-5D-5L) the most used econometric instrument in the world. It is a generic instrument, applicable both in the general population and in patients with different conditions. It contains 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It generates a single score that incorporates society's preferences for health states (utilities), suitable for cost-utility analysis by calculating quality-adjusted life years (QALYs). The health index range from 1 (perfect health) to negative values (for those states considered worse than death), 0 being the value assigned to death. The EQ-5D-5L has been validated in the Spanish population
Changes in quality of life: WHOQOL-BREF | Screening, 6, 12 and 15 months
  Changes in quality of life measured by the the World Health Organization brief generic questionnaire (WHOQOL-BREF), a cross-cultural instrument to assess quality of life. It assesses the following broad domains: physical health, psychological health, social relationships, and environment

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Barcelonabeta Brain Research Center, Barcelona, Barcelona, Spain
  - Hospital del Mar Research Institute Barcelona, Barcelona

REFERENCES:
- [Background] Skaper SD, Facci L, Zusso M, Giusti P. Synaptic Plasticity, Dementia and Alzheimer Disease. CNS Neurol Disord Drug Targets. 2017;16(3):220-233. doi: 10.2174/1871527316666170113120853. PMID 28088900
- [Background] Lopez-Sanz D, Bruna R, Garces P, Martin-Buro MC, Walter S, Delgado ML, Montenegro M, Lopez Higes R, Marcos A, Maestu F. Functional Connectivity Disruption in Subjective Cognitive Decline and Mild Cognitive Impairment: A Common Pattern of Alterations. Front Aging Neurosci. 2017 Apr 21;9:109. doi: 10.3389/fnagi.2017.00109. eCollection 2017. PMID 28484387
- [Background] Mandolesi L, Gelfo F, Serra L, Montuori S, Polverino A, Curcio G, Sorrentino G. Environmental Factors Promoting Neural Plasticity: Insights from Animal and Human Studies. Neural Plast. 2017;2017:7219461. doi: 10.1155/2017/7219461. Epub 2017 Jun 14. PMID 28740740
- [Background] Galvin JE. Prevention of Alzheimer's Disease: Lessons Learned and Applied. J Am Geriatr Soc. 2017 Oct;65(10):2128-2133. doi: 10.1111/jgs.14997. Epub 2017 Aug 2. PMID 28766695
- [Background] De la Torre R, De Sola S, Pons M, Duchon A, de Lagran MM, Farre M, Fito M, Benejam B, Langohr K, Rodriguez J, Pujadas M, Bizot JC, Cuenca A, Janel N, Catuara S, Covas MI, Blehaut H, Herault Y, Delabar JM, Dierssen M. Epigallocatechin-3-gallate, a DYRK1A inhibitor, rescues cognitive deficits in Down syndrome mouse models and in humans. Mol Nutr Food Res. 2014 Feb;58(2):278-88. doi: 10.1002/mnfr.201300325. Epub 2013 Sep 14. PMID 24039182
- [Background] de la Torre R, de Sola S, Hernandez G, Farre M, Pujol J, Rodriguez J, Espadaler JM, Langohr K, Cuenca-Royo A, Principe A, Xicota L, Janel N, Catuara-Solarz S, Sanchez-Benavides G, Blehaut H, Duenas-Espin I, Del Hoyo L, Benejam B, Blanco-Hinojo L, Videla S, Fito M, Delabar JM, Dierssen M; TESDAD study group. Safety and efficacy of cognitive training plus epigallocatechin-3-gallate in young adults with Down's syndrome (TESDAD): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Jul;15(8):801-810. doi: 10.1016/S1474-4422(16)30034-5. PMID 27302362
- [Background] Pons-Espinal M, Martinez de Lagran M, Dierssen M. Environmental enrichment rescues DYRK1A activity and hippocampal adult neurogenesis in TgDyrk1A. Neurobiol Dis. 2013 Dec;60:18-31. doi: 10.1016/j.nbd.2013.08.008. Epub 2013 Aug 20. PMID 23969234
- [Background] Catuara-Solarz S, Espinosa-Carrasco J, Erb I, Langohr K, Notredame C, Gonzalez JR, Dierssen M. Principal Component Analysis of the Effects of Environmental Enrichment and (-)-epigallocatechin-3-gallate on Age-Associated Learning Deficits in a Mouse Model of Down Syndrome. Front Behav Neurosci. 2015 Dec 11;9:330. doi: 10.3389/fnbeh.2015.00330. eCollection 2015. PMID 26696850
- [Background] McEwen SC, Siddarth P, Rahi B, Kim Y, Mui W, Wu P, Emerson ND, Lee J, Greenberg S, Shelton T, Kaiser S, Small GW, Merrill DA. Simultaneous Aerobic Exercise and Memory Training Program in Older Adults with Subjective Memory Impairments. J Alzheimers Dis. 2018;62(2):795-806. doi: 10.3233/JAD-170846. PMID 29480182
- [Background] Prince M, Comas-Herrera A, Knapp M, Guerchet M, Karagiannidou M. World Alzheimer Report 2016 Improving healthcare for people living with dementia. Coverage, Quality and costs now and in the future. Alzheimer's Disease International (ADI). London; 2016.
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Buckley RF, Maruff P, Ames D, Bourgeat P, Martins RN, Masters CL, Rainey-Smith S, Lautenschlager N, Rowe CC, Savage G, Villemagne VL, Ellis KA; AIBL study. Subjective memory decline predicts greater rates of clinical progression in preclinical Alzheimer's disease. Alzheimers Dement. 2016 Jul;12(7):796-804. doi: 10.1016/j.jalz.2015.12.013. Epub 2016 Feb 4. PMID 26852195
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Crous-Bou M, Minguillon C, Gramunt N, Molinuevo JL. Alzheimer's disease prevention: from risk factors to early intervention. Alzheimers Res Ther. 2017 Sep 12;9(1):71. doi: 10.1186/s13195-017-0297-z. PMID 28899416
- [Background] Vellas B, Carrie I, Gillette-Guyonnet S, Touchon J, Dantoine T, Dartigues JF, Cuffi MN, Bordes S, Gasnier Y, Robert P, Bories L, Rouaud O, Desclaux F, Sudres K, Bonnefoy M, Pesce A, Dufouil C, Lehericy S, Chupin M, Mangin JF, Payoux P, Adel D, Legrand P, Catheline D, Kanony C, Zaim M, Molinier L, Costa N, Delrieu J, Voisin T, Faisant C, Lala F, Nourhashemi F, Rolland Y, Van Kan GA, Dupuy C, Cantet C, Cestac P, Belleville S, Willis S, Cesari M, Weiner MW, Soto ME, Ousset PJ, Andrieu S. MAPT STUDY: A MULTIDOMAIN APPROACH FOR PREVENTING ALZHEIMER'S DISEASE: DESIGN AND BASELINE DATA. J Prev Alzheimers Dis. 2014 Jun;1(1):13-22. PMID 26594639
- [Background] Andrieu S, Guyonnet S, Coley N, Cantet C, Bonnefoy M, Bordes S, Bories L, Cufi MN, Dantoine T, Dartigues JF, Desclaux F, Gabelle A, Gasnier Y, Pesce A, Sudres K, Touchon J, Robert P, Rouaud O, Legrand P, Payoux P, Caubere JP, Weiner M, Carrie I, Ousset PJ, Vellas B; MAPT Study Group. Effect of long-term omega 3 polyunsaturated fatty acid supplementation with or without multidomain intervention on cognitive function in elderly adults with memory complaints (MAPT): a randomised, placebo-controlled trial. Lancet Neurol. 2017 May;16(5):377-389. doi: 10.1016/S1474-4422(17)30040-6. Epub 2017 Mar 27. PMID 28359749
- [Background] Moll van Charante EP, Richard E, Eurelings LS, van Dalen JW, Ligthart SA, van Bussel EF, Hoevenaar-Blom MP, Vermeulen M, van Gool WA. Effectiveness of a 6-year multidomain vascular care intervention to prevent dementia (preDIVA): a cluster-randomised controlled trial. Lancet. 2016 Aug 20;388(10046):797-805. doi: 10.1016/S0140-6736(16)30950-3. Epub 2016 Jul 26. PMID 27474376
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Valls-Pedret C, Lamuela-Raventos RM, Medina-Remon A, Quintana M, Corella D, Pinto X, Martinez-Gonzalez MA, Estruch R, Ros E. Polyphenol-rich foods in the Mediterranean diet are associated with better cognitive function in elderly subjects at high cardiovascular risk. J Alzheimers Dis. 2012;29(4):773-82. doi: 10.3233/JAD-2012-111799. PMID 22349682
- [Background] Martinez-Lapiscina EH, Clavero P, Toledo E, San Julian B, Sanchez-Tainta A, Corella D, Lamuela-Raventos RM, Martinez JA, Martinez-Gonzalez MA. Virgin olive oil supplementation and long-term cognition: the PREDIMED-NAVARRA randomized, trial. J Nutr Health Aging. 2013;17(6):544-52. doi: 10.1007/s12603-013-0027-6. PMID 23732551
- [Background] Valls-Pedret C, Sala-Vila A, Serra-Mir M, Corella D, de la Torre R, Martinez-Gonzalez MA, Martinez-Lapiscina EH, Fito M, Perez-Heras A, Salas-Salvado J, Estruch R, Ros E. Mediterranean Diet and Age-Related Cognitive Decline: A Randomized Clinical Trial. JAMA Intern Med. 2015 Jul;175(7):1094-1103. doi: 10.1001/jamainternmed.2015.1668. PMID 25961184
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666